CLINICAL TRIAL: NCT00741858
Title: Prospective Randomized Study of Duragen vs. Duraguard in Chiari Surgery
Brief Title: Duragen Versus Duraguard in Chiari Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Konstantin V. Slavin, Professor Neurologic Surgery, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIC 2002-0232; NCT00565435 (obsolete NCT alias)
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Chiari Malformation
Keywords: Chiari malformation;; Duraplasty;; Posterior fossa decompression;; Duragen;; Duraguard
MeSH Terms: conditions — Arnold-Chiari Malformation | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DuraGen (sutureless) (Experimental): Duragen duraplasty - the Duragen patch is applied over the dural defect during Chiari decompression surgery. The Duragen represents sutureless technique of posterior fossa duraplasty. Rest of the treatment is as usual.
  Interventions: Procedure: Duragen duraplasty
- DuraGuard (suturable) (Active Comparator): Duraguard duraplasty - the Duraguard patch is applied over the dural defect during Chiari decompression surgery and sutured to the dural edge. This represents suturable technique that theoretically provides better (water-tight) dural closure.
  Interventions: Procedure: Duraguard duraplasty

INTERVENTIONS:
Procedure: Duragen duraplasty — Posterior cranial fossa repair and enlargement with application of dural patch (Duragen)
  Other Names: Duragen (Arm 1; active comparator)
  Arms: DuraGen (sutureless)
Procedure: Duraguard duraplasty — Posterior cranial fossa repair and enlargement with application of dural patch (Duraguard)
  Other Names: Duraguard (Arm 2; active comparator)
  Arms: DuraGuard (suturable)

SUMMARY:
The study evaluates two materials used for duraplasty of the posterior cranial fossa in treatment of Chiari malformation. One material (DuraGen) is a non-suturable collagen matrix that is applied over the defect if brain coverings (dura); the other (DuraGuard) is made out of bovine pericardium and has to be sutured during application. The study compares these two materials used for duraplasty of patients undergoing Chiari surgery in a prospective randomized fashion to check the rate of surgical complications associated with each material, patient's outcomes, length of surgery and the hospital stay, etc.

DETAILED DESCRIPTION:
The study is aimed at comparative analysis of two frequently used duraplasty materials: one is made out of bovine pericardium, and the other - from bovine collagen derived from bovine achilles tendon. Both materials are routinely used form this intervention (duraplasty), but the question of superiority of one over the other remains open. This study follows patients with Chiari malformation from the time of surgery to the time of their discharge from the hospital and then another 3 months of follow up care.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Chiari malformation

Exclusion Criteria:

* Presence of ventriculoperitoneal shunt
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-04; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin V Slavin, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center in Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: Departmental website — http://chicago.medicine.uic.edu/departments___programs/departments/neurosurgery/

RESULTS

PARTICIPANT FLOW:
Groups:
- DuraGen (Sutureless): Duragen - the Duragen patch is applied over the dural defect during Chiari decompression surgery. The Duragen represents sutureless technique of posterior fossa duraplasty. Rest of the treatment is as usual.
  Duraplasty with Duragen: Posterior cranial fossa repair and enlargement with application of dural patch (Duragen)
- DuraGuard (Suturable): Duraguard - the Duraguard patch is applied over the dural defect during Chiari decompression surgery and sutured to the dural edge. This represents suturable technique that theoretically provides better (water-tight) dural closure.
  Duraplasty with Duraguard: Posterior cranial fossa repair and enlargement with application of dural patch (Duraguard)
Period: Overall Study
Arm/Group | DuraGen (Sutureless) | DuraGuard (Suturable)
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DuraGen (Sutureless) | DuraGuard (Suturable) | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12) | 39 (12) | 38.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Physical Health Quality of Life
Description: Physical health quality of life (based on SF-36 results) (SF-36 includes 8 scores scaled 0-100; lower score indicating more disability)
Time Frame: 7 years
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DuraGen (Sutureless) | DuraGuard (Suturable)
Number analyzed (Participants) | 16 | 18
units on a scale | 31.4 (2.01) | 35.61 (1.87)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | DuraGen (Sutureless) | DuraGuard (Suturable)
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/18
Other Adverse Events (participants affected / at risk) | 1/16 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DuraGen (Sutureless) (N=16) | DuraGuard (Suturable) (N=18)
CSF leak (Nervous system disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DuraGen (Sutureless) (N=16) | DuraGuard (Suturable) (N=18)
meningitis (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No